CLINICAL TRIAL: NCT00962481
Title: A Double-blind, Placebo Controlled, Randomized, Cross-over, Phase IIa Study to Evaluate the Effect of Bimosiamose on Ozone Induced Sputum Neutrophilia in Healthy Subjects
Brief Title: Study to Evaluate the Effect of Bimosiamose on Ozone Induced Sputum Neutrophilia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revotar Biopharmaceuticals AG (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R014
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — bimosiamose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Bimosiamose (Active Comparator)
  Interventions: Drug: Bimosiamose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bimosiamose
  Arms: Bimosiamose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of repeated inhalative doses of Bimosiamose on ozone induced sputum neutrophilia in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to produce sputum with normal sputum neutrophil levels at screening (< 65% of non-epithelial cells).
* Ozone responsive, defined as ≥ 20% relative increase in sputum neutrophils cell count after 3 h ozone challenge.
* At screening FEV1 at least 80% of predicted.

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 3 months). Urine cotinine levels will be measured during screening for all subjects. Smokers will be defined as any subject who reports of a recent tobacco use and/or who has a urine cotinine ≥ 500 ng/mL.
* Significant illness within two weeks prior to dosing (e.g., infection).
* Recent (within the last three years) and/or recurrent history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Pneumologisches Forschungsinstitut GmbH am Krankenhaus Großhansdorf, Großhansdorf, Germany